CLINICAL TRIAL: NCT01620567
Title: The Effect of Consumption of Potatoes, Avocados and Chickpeas Daily for 6 Months on Cognitive Function in Older Adults
Brief Title: Consumption of Potatoes, Avocados and Chickpeas and Cognitive Function in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 002
Record Dates: First submitted 2012-06-13; First posted 2012-06-15 (Estimated); Results first posted 2019-07-19 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-05

CONDITIONS: Mild Cognitive Impairment
Keywords: lutein; avocados; chickpeas; potatoes; elderly
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- chickpeas/potatoes (Placebo Comparator): 1 potato/day or 1 cup chickpeas
  Interventions: Other: potato or chickpea
- avocados (Active Comparator): 1 avocados/day
  Interventions: Other: avocado

INTERVENTIONS:
Other: avocado — 1 avocado/day for 6 months
  Arms: avocados
Other: potato or chickpea — 1 cup potatoes or chickpeas/day for 6 months
  Arms: chickpeas/potatoes

SUMMARY:
Cognitive impairment is also a major risk factor for development of dementia later in life. Findings from the investigators studies suggest that the carotenoids, lutein and zeaxanthin may be important in cognitive function in the elderly. Avocados are a source of these carotenoids. The investigators study evaluates long-term avocado intervention as a treatment strategy for age-related cognitive impairment which could possibly prevent the onset of dementia. The investigators have also shown that lutein supplementation significantly improved verbal fluency scores in healthy older women. Based on these findings, the next logical step will be to investigate the ability of lutein and zeaxanthin contained in avocados to influence cognitive function in older adults. The investigators hypothesize that there will be a significant increase in cognitive function measures in older adults provided with meals containing 1 avocado/day at the end of 6 months, while no significant improvements will be observed in older adults given daily meals containing chickpeas and/or potatoes.

The proposed study is designed as a randomized, placebo controlled trial that tests the effects of 6 month supplementation with 1 avocado/day on cognitive function in older adults. Secondary analyses will determine whether baseline macular pigment (lutein in retina which canbe measured non invasivley) density predicts relative effectiveness of the intervention on cognitive function. Secondary outcomes include plasma biomarkers of oxidative stress and inflammation.

DETAILED DESCRIPTION:
The study is designed as a placebo controlled trial that tests the effects of 6 month supplementation with daily meals containing 1 avocado or isocaloric amounts of chickpeas and/or potatoes on cognitive function in older adults. Subjects will be randomly assigned to one of the two groups. Secondary analyses will determine whether baseline macular pigment density (a non invasive measure of lutein and zeaxanthin in neural tissue) predicts relative effectiveness of the intervention on cognitive function. Secondary outcomes include plasma biomarkers of oxidative stress and inflammation. Participants will be recruited from community-dwelling men and women aged >50 yr, and potential participants will be screened to meet cognitive and functional criteria. Participants will be pre-screened by telephone; those who appear to meet criteria will undergo further screening. The study will include baseline (0 month), 3 and 6 month visits for study procedures, and monthly telephone calls. Given that there is a visible difference between the two interventions, a blinded study is not possible.

ELIGIBILITY:
Inclusion Criteria:

* men and women age > 50 years
* BMI 19-30 kg/m2
* lutein intake of < 3 mg/d
* Docosahexaenoic acid intake < 250 mg/d (including supplements)
* Mini mental state exam (MMSE) score > 24
* Macular pigment density < 0.4 at 0.5 degrees
* Beck Depression Inventory < 20
* free of known disease
* BMI 19-29 kg/m2
* must be able to give written informed consent
* have normal hematologic parameters
* normal values of plasma albumin
* normal values for liver and kidney function (Appendix A)
* no use of carotenoid, n3 fatty acid, multivitamin/mineral, (> 2 months).

Exclusion Criteria:

* history of active small bowel disease or resection
* atrophic gastritis
* hyperlipidemia (LDL >120 mg/dL or triglycerides >150 mg/dL)
* hypertension (>150/90 mm Hg)
* diabetes, alcoholism (>2 drinks/d or 14 drinks/week)
* pancreatic disease
* anemia, and bleeding disorders (as determined by screening interview)
* avocado, potato or chickpea allergy
* pregnancy or lactation
* diseases that interfere with fat absorption, e.g. colitis, celiac disease, Crohn's disease, cystic fibroids (as determined by screening interview)
* medications that interfere with fat absorption, e.g. bile sequestrants (as determined by screening interview)
* use of antipsychotic, antimanic, anti-inflammatory, monoamine inhibitors, or dementia medications
* smoking or use of nicotine patches or gum (within past 6 months)
* use of drugs suspected of interfering with metabolism of blood clotting, e.g. warfarin (as determined by screening interview)
* subjects having extremely high dietary intakes of carotenoids as indicated by screening plasma values > NHANES 95th percentile for lutein/zeaxanthin, beta-carotene, cryptoxanthin, or lycopene
* stroke,head injury with loss of consciousness or seizures.
* Non English speaking: This is a small study with a sample size. Logistically and financially, getting materials translated for such a small study is not feasible.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth J Johnson, Ph.D., Principal Investigator — Tufts University
Locations (1):
- Jean Mayer USDA Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Chickpeas/Potatoes: 1 cup of chickpeas/potatoes for 6 months
- Avocados: 1 avocado/day for 6 months
Period: Overall Study
Arm/Group | Chickpeas/Potatoes | Avocados
Started | 23 | 25
Completed | 20 | 20
Not Completed | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Chickpeas/Potatoes: 1 cup chickpeas/potatoes for 6 months
- Total: Total of all reporting groups
Arm/Group | Chickpeas/Potatoes | Avocados | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 12 | 27
  >=65 years | 5 | 8 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 9 | 7 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 14 | 13 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Cognition
Description: measures of sustained attention will be made using CANTAB, a sensitive computerized program. Signal detection measured on a scale from 0 to 1(bad to good).
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Chickpeas/Potatoes: 1 potato/day or 1 cup chickpeas for 6 months
Arm/Group | Chickpeas/Potatoes | Avocados
Number analyzed (Participants) | 20 | 20
units on a scale
  baseline - rapid visual information processing | .90 (.05) | .86 (.21)
  3 mo - rapid visual information processing | .92 (.05) | .92 (.04)
  6 mo - rapid visual information processing | .92 (.05) | .93 (.04)

2. Secondary Outcome: Inflammation
Description: C-reactive protein
Time Frame: 0 months
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Chickpeas/Potatoes | Avocados
Number analyzed (Participants) | 20 | 20
mg/L | 1.3 (1.0) | 2.0 (2.8)

3. Secondary Outcome: Inflammation
Description: C-reactive protein
Time Frame: 3 month
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Chickpeas/Potatoes | Avocados
Number analyzed (Participants) | 20 | 20
mg/L | 2.3 (2.4) | 2.0 (2.8)

4. Secondary Outcome: Inflammation
Description: C-reactive protein
Time Frame: 6 month
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Chickpeas/Potatoes | Avocados
Number analyzed (Participants) | 20 | 20
mg/L | 1.6 (1.6) | 1.7 (1.8)

ADVERSE EVENTS:
Groups:
- Avocados: avocados
  1 avocado/day for 6 months
Arm/Group | Chickpeas/Potatoes | Avocados
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/25
Other Adverse Events (participants affected / at risk) | 0/23 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No